CLINICAL TRIAL: NCT01377168
Title: Oral Naltrexone for Improved Medication Compliance Among HIV-infected Men With Alcohol Use Disorder
Brief Title: Naltrexone for Medication Compliance Among HIV-infected Men With Alcohol Use Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Yale University (Other); Asociación Civil Impacta Salud y Educación, Peru (Other)
Responsible Party: Principal Investigator, Ann C Duerr, Member, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XR-NTX ETOH
Record Dates: First submitted 2011-06-17; First posted 2011-06-21 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: HIV; Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo pill (Placebo Comparator): Daily oral placebo.
  Interventions: Drug: Placebo pill
- NTX (Active Comparator): Daily oral naltrexone.
  Interventions: Drug: oral naltrexone

INTERVENTIONS:
Drug: oral naltrexone
  Other Names: Nalerona
  Arms: NTX
Drug: Placebo pill
  Arms: Placebo pill

SUMMARY:
This study will recruit 159 HIV-infected men with alcohol use disorders (AUDs). Men will be randomized to receive either oral naltrexone for the treatment of alcohol use disorder or placebo. Men with acute, recent or established HIV infection will receive antiretroviral treatment (ART) and be randomized to oral naltrexone or placebo. The purpose of this study is to see whether use of oral naltrexone improves medication compliance, and therefore HIV viral load suppression, among men with alcohol use disorder. The study will also assess the impact of oral naltrexone on alcohol use behaviors in this population.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for alcohol dependence or problem drinking.
* Age 18 years and older
* Confirmed HIV infection, either through positive HIV antibody or detectable HIV-1 RNA level.
* No participation in pharmacotherapy trial in the previous 30 days
* Not pregnant

Exclusion Criteria:

* Unable to provide informed consent
* Verbally or physically threatening to research staff
* Unable to communicate in Spanish
* Pending trials for a felony
* Childs-Pugh Class C Cirrhosis
* Grade 3 Hepatitis (LFTs > 5X normal)
* Receiving opioid prescription narcotics or has pain syndrome necessitating future use of opioid prescription narcotics.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2014-05; Primary Completion 2016-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
HIV Viral Load Suppression | 6 months
  The primary outcome will be the proportion with a VL<400 copies/mL at 6 months.

SECONDARY OUTCOMES:
ART Compliance and Alcohol Use Behavior | 6 months
  Secondary HIV outcomes will include time to ART initiation, retention on ART over 6 months, and HIV sexual risk behaviors. Alcohol use outcomes include the following: 1) Time to relapse to heavy drinking (for men defined as >5 drinks/drinking day); 2) percent of days drinking (PDD) over the six-month examination period; 3) percent of days abstinent (PDA) over the six month examination period; and 4) alcohol craving using the Obsessive Compulsive Drinking Scale where a mean change in total score will be assessed and compared between treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Duerr, MD, PhD, MPH, Principal Investigator — Fred Hutchinson Cancer Center; Frederick Altice, MD, Study Director — Yale University
Locations (1):
- Asociación Civil Impacta Salud y Educación, Lima, Peru